CLINICAL TRIAL: NCT02712593
Title: A Randomized, Double-blind, Placebo Controlled Parallel Study Investigating the Effects of Niagen™ (Nicotinamide Riboside) on Niagen™ Metabolites in Healthy Adults.
Brief Title: A Study Investigating the Effects of Niagen™ in Healthy Adults.
Acronym: 15NRHC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KGK Science Inc. (Industry)
Collaborators: ChromaDex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 15NRHC
Record Dates: First submitted 2016-03-01; First posted 2016-03-18 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Bioavailability
Keywords: Healthy participants; Dietary supplement; Bioavailability; Niagen™; Nicotinamide riboside; N-methylnicotinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Niagen™ 100 (Experimental)
  Interventions: Dietary Supplement: Niagen™ 100
- Niagen™ 300 (Experimental)
  Interventions: Dietary Supplement: Niagen™ 300
- Niagen™ 1000 (Experimental)
  Interventions: Dietary Supplement: Niagen™ 1000
- Placebo (Experimental)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Niagen™ 100
  Arms: Niagen™ 100
Dietary Supplement: Niagen™ 300
  Arms: Niagen™ 300
Dietary Supplement: Niagen™ 1000
  Arms: Niagen™ 1000
Other: Placebo
  Arms: Placebo

SUMMARY:
This study will evaluate the effect of repeated doses of Niagen™ on Niagen™ metabolite concentrations in blood, urine and muscle. There will be 3 doses of Niagen™ compared to a placebo. One quarter of subjects will receive the low dose of Niagen™, one quarter will receive the moderate dose of Niagen™, one quarter will receive the higher dose of Niagen™ and one quarter will reveive the placebo.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25-30kg/m²
* If female, subject is not of child bearing potential, which is defined as females who have had a hysterectomy or oophorectomy, bilateral tubal ligation or are post-menopausal (natural or surgically with > 1 year since last menstruation) OR Females of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result. Acceptable methods of birth control include:

  * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
  * Double-barrier method
  * Non-hormonal intrauterine devices
  * Vasectomy of partner
* Healthy as determined by laboratory results, medical history, and physical exam
* Agrees to comply with study procedure
* Agrees to maintain current level of physical activity throughout the study and avoid exercising on the day of study visits 3 to 7 (prior to the visit).
* Agrees to refrain from consuming caffeine (i.e. coffee) on the days of study visits 3 to 7 (prior to the visit)
* Agrees to avoid taking Vitamin B3 (niacin, nicotinic acid,niacinamide) supplements or multivitamins 14 days prior to randomization and for the duration of the study period
* Has given voluntary, written, informed consent to participate in the study
* Agrees to avoid foods that contain high amounts of tryptophan and niacin and limit their ingestion of foods containing moderate amounts of tryptophan and niacin

Exclusion Criteria:

* Women who are pregnant, breastfeeding, or planning to become pregnant during the course of the trial
* Alcohol use >2 standard alcoholic drinks per day
* History of alcohol or drug abuse within the past year
* Medicinal use of marijuana
* Diabetes (Type I or Type II)
* Subjects taking lipid lowering drugs
* History of renal and/or liver disease
* History of pellagra or niacin deficiency
* Significant or untreated medical disorders including recent myocardial ischemia or infarction, unstable angina, uncontrolled hypertension, AIDS, malignancy, and neurological disorders including epilepsy, and recent cerebrovascular disease
* Subjects with or who had recently experienced a traumatic injury, inflammation, infections or had undergone surgery
* Use of natural health products containing NR within 14 days prior to randomization and during the course of the study
* Unstable medical conditions as determined by the Qualified Investigator
* Clinically significant abnormal lab results at screening (e.g. AST and/or ALT > 2 x ULN, and/or bilirubin > 2 x ULN) will be assessed by the Medical Investigator
* History of or current diagnosis of any cancer (except for successfully treated basal cell carcinoma) diagnosed less than 5 years prior to screening. Subjects with cancer in full remission more than 5 years after diagnosis are acceptable
* Participation in a clinical research trial within 30 days prior to randomization
* Allergy or sensitivity to study supplement ingredients
* Allergy or sensitivity to lidocaine
* Bleeding disorder
* Serum creatinine ≥ 130µmol/L for males and ≥ 125µmol/L for female
* Individuals who are cognitively impaired and/or who are unable to give informed consent
* Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or which may pose significant risk to the subjects

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2016-03-21 (Actual); Primary Completion 2017-03-17 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Urinary Methylnicotinamide | 8 weeks: from baseline to end of study
  Change in levels

SECONDARY OUTCOMES:
Blood Nicotinamide Riboside Metabolites | 8 weeks: from baseline to end of study
  Change in levels
Urinary Nicotinamide Riboside Metabolites | 8 weeks: from baseline to end of study
  Change in levels
Muscle Nicotinamide Riboside Metabolites | 8 weeks: from baseline to end of study
  Change in Levels of Metabolites Assessed from Muscle Tissue collected with Micro-Needle Biopsy

OTHER OUTCOMES:
Resting Metabolic Rate | 8 weeks: from baseline to end of study
  Change in Levels (kcal/day) Assessed by the ReeVue Indirect Calorimeter
Expression profile: Branched Amino Acids | 8 weeks: from baseline to end of study
Expression profile: high sensitivity C-reactive protein | 8 weeks: from baseline to end of study
Incidence of Abnormal Vital Signs | 8 weeks: from baseline to end of study
  Resting blood pressure
Incidence of Abnormal Laboratory Values | 8 weeks: baseline to end of study
  Assessment of hematology and clinical chemistry parameters: CBC, electrolytes (Na, K, CL), AST, ALT, GGT, BUN, HDL, LDL, triglycerides and total cholesterol
Incidence of Adverse Events | 8 weeks: baseline to end of study
  Review of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Schacter, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Synergize Inc., London, Ontario, Canada